CLINICAL TRIAL: NCT04246164
Title: A Randomized, Double-Blinded, Placebo Controlled Pilot Trial of the Feasibility of High Definition Transcranial Direct Current Stimulation and Cognitive Training in Patients With Mild Cognitive Impairment.
Brief Title: A Study of HD-tDCS and Cognitive Training to Improve Cognitive Function in MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Priyanka Shah-Basak, PhD, Assistant Professor of Neurology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00035757
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Memory Disorders; Memory Loss
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Intervention Model Description: placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HD-tDCS combined with CT (Active Comparator): HD-tDCS combined with CT, administered to participants with amnestic MCI (aMCI) in blocks of 5 daily treatments for a total of 15 sessions. There will be one treatment block/month for a total of 3 months
  Interventions: Device: HD-tDCS combined with CT
- sham HD-tDCS combined with CT (Sham Comparator): sham HD-tDCS combined with CT, administered to participants with amnestic MCI (aMCI) in blocks of 5 daily treatments for a total of 15 sessions. There will be one treatment block/month for a total of 3 months
  Interventions: Device: sham HD-tDCS combined with CT

INTERVENTIONS:
Device: HD-tDCS combined with CT — HD-tDCS treatments will be administered during a cognitive training session.
  Arms: HD-tDCS combined with CT
Device: sham HD-tDCS combined with CT — sham-HD-tDCS treatments will be administered during a cognitive training session.
  Arms: sham HD-tDCS combined with CT

SUMMARY:
The primary objective of this project is to assess the feasibility of multi-field, extended HD-tDCS (MFE-HD-tDCS) with simultaneous computerized CT as a viable intervention to improve cognitive function in patients with MCI. This double-blinded, randomized pilot clinical trial of repetitive daily HD-tDCS/sham HD-tDCS, administered in combination with CT to subjects with MCI in 3 monthly blocks of 5 daily sessions for a total of 15 sessions will enroll 8 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50-90 years
2. Willing and able to undergo all procedures
3. Retains decisional capacity at initial visit
4. Meets criteria for MCI, amnestic type (Petersen, 2004).

Exclusion Criteria:

1. Significant kidney injury requiring hemodialysis
2. Automatic Internal Cardiac Defibrillator (AICD) or Pacemaker
3. Significant congestive heart failure
4. History of clinically significant ischemic or hemorrhagic stroke, or lacune or infarct considered by radiologist likely to cause or contribute significantly to cognitive symptoms
5. History of thalamic lacunar stroke
6. Modified Hachinski Ischemia Score >4 points
7. History of seizure disorder requiring medication
8. History of brain surgery (for seizure disorder, aneurysms, or benign/malignant tumor)
9. History of HIV/AIDS
10. Severe untreated obstructive sleep apnea
11. Greater than three servings alcohol daily or illicit drug use
12. Major neurologic disorders other than dementia (e.g., MS, ALS)
13. Schizophrenia, bipolar disorder, other serious mental illnesses
14. Other significant medical conditions at investigators' discretion
15. Pregnancy
16. Lack of study partner (Participants are allowed to find a new study partner if the original study partner withdraws)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject signed the consent form and withdrew prior to being assigned to one of the treatment arms.
Period: Overall Study
Arm/Group | HD-tDCS Combined With CT | Sham HD-tDCS Combined With CT
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HD-tDCS Combined With CT | Sham HD-tDCS Combined With CT | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Assess the Feasibility of MFE-HD-tDCS Plus Simultaneous Computerized CT as a Viable Intervention by Measuring Consent Rates and Treatment Completion
Description: This measure assesses consent rates and treatment completion amongst subjects by assessing the number of subjects who signed consent forms and the number of completed study visits.
  In this study, 9 subjects provided informed consent. 1 subject was withdrawn. 8 subjects completed treatment. Therefore, only the data from the 8 subjects who completed treatment were analyzed.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HD-tDCS Combined With CT | Sham HD-tDCS Combined With CT
Number analyzed (Participants) | 4 | 4
Participants
  Number of subjects who signed consent forms | 4 | 4
  Number of subjects who completed study treatment | 4 | 4

2. Secondary Outcome: Collect Preliminary Data on the Efficacy of MFE-HD-tDCS With Simultaneous Computerized CT
Description: Alzheimer's Disease Cooperative Study Preclinical Alzheimer Cognitive Composite (ADCS-PACC) is a composite of 4 measures with well-established sensitivity for the detection of cognitive decline in prodromal and mild dementia. It is calculated by summing the standardized z-scores of each of the following:
  * Rey Auditory Verbal Learning Test (0-48 points), Logical Memory IIa sub-test from the Wechsler Memory test (0-25 points)
  * Mini Mental Status Examination (0-30 points)
  * Digit Symbol Substitution Test from the Wechsler Adult Intelligence Scale-Revised (0-93 points)
  Z-score of 0 represents the sample mean. A Z-score of 0 indicates average cognitive performance compared to the reference group.
  For ADCS-PACC, more standard deviations above the mean generally represent a better outcome.
  There are not specific clinically relevant thresholds universally agreed upon for ADCS-PACC scores. Scores are typically used to compare changes over time.
Time Frame: Alzheimer's Disease Cooperative Study, Preclinical Alzheimer's Cognitive Composite (ADCS-PACC) score at 3 and 6 months from baseline.
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | HD-tDCS Combined With CT | Sham HD-tDCS Combined With CT
Number analyzed (Participants) | 4 | 4
Z-Score
  Mean ADCS-PACC at Baseline | -0.95975 (2.2504557131094) | 0.85375 (3.3297438715313)
  Mean ADCS-PACC at Month 3 | -0.795 (2.5196990561044) | 1.596 (3.2651291960146)
  Mean ADCS-PACC at Month 6 | -0.38575 (3.5756851441367) | 1.227 (2.764333011777)

3. Secondary Outcome: Collect Preliminary Data on the Efficacy of MFE-HD-tDCS in Combination With Computerized CT to Improve Quality of Life in Subjects With MCI
Time Frame: Measure quality of life in subjects over a period of 3 months
Population: Quality of life questionnaires were removed from study procedures prior to subject enrollment. Therefore, we did not have adequate data to support this outcome measure, so no data is reported. For this reason, no statistical analysis was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | HD-tDCS Combined With CT | Sham HD-tDCS Combined With CT
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

4. Secondary Outcome: Effects of MFE-HD-tDCS Combined With Computerized CT on Resting State Brain Network Connectivity
Description: To report the correlation between activation in different brain regions reported.
  The clinical significance of increasing or reducing connectivity remains unclear. For example, increased connectivity could lead to strengthening of a hypo-functioning network, but reducing connectivity could also be the result of normalizing aberrant and/or compensatory hypo-connectivity.
  Calculation details:
  Pearson r correlation coefficients were computed and transformed to Fisher-z. Independent t-test or Wilcoxon Rank Sum analyses were conducted to investigate changes in connectivity from pre- to post-intervention between groups (Active versus Sham).
  Higher Z-scores (standard deviations above the mean) represent greater functional connectivity (stronger temporal synchronization) between the specified regions of interest (ROIs). Lower Z-scores represent reduced functional connectivity (weaker synchronization).
  A decrease in Z-scores (lower connectivity) is considered a better outcome.
Time Frame: 3 months
Population: We analyzed resting state connectivity changes at Month 3 on MRI
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | HD-tDCS Combined With CT | Sham HD-tDCS Combined With CT
Number analyzed (Participants) | 4 | 4
Z-score
  Resting state connectivity changes between left caudal hippocampus and left lateral parietal cortex | -0.09065 (0.018280796) | 0.12688 (0.046184866)
  Resting state connectivity changes between right intraparietal sulcus and right frontal eye fields | -0.0989 (0.081790097) | 0.11118 (0.046729989)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored recorded from the time of informed consent through study completion, an average of 6 months per subject.
Arm/Group | HD-tDCS Combined With CT | Sham HD-tDCS Combined With CT
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD-tDCS Combined With CT (N=4) | Sham HD-tDCS Combined With CT (N=4)
Gallbladder removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Gall stones (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD-tDCS Combined With CT (N=4) | Sham HD-tDCS Combined With CT (N=4)
Common cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT04246164/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT04246164/ICF_001.pdf